CLINICAL TRIAL: NCT05204576
Title: Computer Based Treatment for Cognitive Behavioral Therapy and Cooperative Pain Education and Self-Management
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000026276; 1R61AT010619-01 (NIH); 4R33AT010619-02 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2022-01-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Chronic Pain
Keywords: Opioid-use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care treatment as usual (TAU) (No Intervention): Individuals will receive buprenorphine or methadone in addition to regular individual or group sessions as offered by the clinic
- CBT4CBT-Copes (Experimental): Individuals will receive standard agonist treatment plus access to the CBT4CBT-COPES website plus daily texts with a link to a survey.
  Interventions: Behavioral: CBT4CBT COPES

INTERVENTIONS:
Behavioral: CBT4CBT COPES — Individuals will receive standard agonist treatment plus access to the CBT4CBT-COPES website plus daily IVR assessment calls
  Arms: CBT4CBT-Copes

SUMMARY:
The investigators plan to develop and pilot test an integrated, web-based cognitive behavioral approach and then conduct a randomized clinical trial evaluating its efficacy relative to standard care in a large and diverse sample of individuals with chronic pain treated with buprenorphine or methadone. The new program will retain key components of Dr. Carroll's computer-based training for cognitive-behavioral therapy (CBT4CBT), including its emphasis on teaching cognitive and behavioral coping skills in an engaging way and focus on the 5 A's of MAT (Adherence, Attendance, Abstinence, Alternate Activities and Accessing support); it will add components from Dr. Heapy's COPES (Cooperative Pain Education and Self-Management) intervention (self-management of chronic pain, with daily surveys via text that monitor pain intensity and interference, physical activity, and skills practice) and modify existing CBT4CBT modules to address the complex interplay between pain and drug use in this population, emphasizing the development of generalizable skills. A randomized clinical trial evaluating CBT4CBT-COPES will be conducted in a diverse sample 160 of individuals enrolled in agonist treatment (methadone or buprenorphine) who have chronic pain, in a 3-month randomized clinical trial with a 6-month follow-up, comparing it to standard treatment alone. The primary retention outcome will be adherence with agonist treatment; the primary pain outcome will be the PROMIS 6-item Pain Interference Short Form.

DETAILED DESCRIPTION:
Evaluate the efficacy of CBT4CBT-COPES versus standard care (treatment as usual) at 3 months (primary endpoint) among 160 individuals with OUD and chronic pain enrolled in OAT at the Liberation clinics. The primary outcome will be adherence to OAT (defined as continuous and verified enrollment at the 3-month timepoint); the primary pain outcome will be pain interference as measured by the PROMIS 6-item Pain Interference Short Form. Hypothesis 1a: Individuals randomized to CBT4CBT-COPES will have greater retention at the 3-month point than those assigned to standard care. Hypothesis 1b: CBT4CBT-COPES will be associated with greater reductions in pain interference at the 3-month point.

2. Conduct a 6-month follow-up to evaluate the durability of effects on the primary outcomes. The investigators hypothesizes CBT4CBT-COPES will be associated with greater adherence and reduced pain interference compared with standard care at the 3 and 6-month follow-ups (6 and 9 months post randomization).

Procedures Initial Screening by Project Manager or Research Assistant: Individuals enrolled in the buprenorphine or methadone programs at Liberation will be informed of the study via flyers, group meetings, or their clinicians. Individuals who indicate they are interested in hearing more about the study will be offered a meeting with the research staff. At the first interview, the research staff will provide an overview of the study and obtain written informed consent. The investigators use a multiple-choice test to assess participants' comprehension of the protocol, with ample time to review questions to assure understanding of the protocol, consent, and treatments offered. After determination of eligibility and informed consent, pre-treatment assessments will be completed. Randomization will occur as soon as participants have achieved a therapeutic dose of buprenorphine or methadone.

Urn randomization. To increase the likelihood that treatment groups are balanced with respect to demographic variables (gender, race), as well as likely prognostic variables (severity of opioid use disorder as moderate or severe via DSM-5 OUD symptom count, initial opioid experience of heroin versus prescription opioids, buprenorphine versus methadone treatment, pain severity (mild, moderate vs. severe) as operationalized by NRS average weekly pain rating). Participants will be assigned to treatment conditions through urn randomization using a Microsoft Access program developed and implemented successfully in multiple previous trials.

Treatment phase: Treatment conditions are described in detail below. Study treatments will last 12 weeks. During the treatment phase, all participants will meet weekly with the research assistant for completion of self-report and interview assessments preferably in-person, but with the option of virtual meetings. Breath and urine sample collection will be taken by the research assistant at this time.

Clinical deterioration: The investigators will closely monitor participant treatment response and safety in all conditions through weekly assessment sessions that will include brief assessment of psychiatric status. Although in the investigators experience this is a very rare event, including during computer-assisted therapy, participants who show significant deterioration (e.g., increased drug/alcohol use or psychiatric symptoms that cannot be managed within the protocol, including significant suicidal or homicidal ideation) will be regarded as symptomatic failures, withdrawn from the treatment arm of the study, and referred for appropriate treatment (usually inpatient care). The project psychiatrist (Dr. Sofuoglu) will make the final withdrawal determination, using guidelines the investigators have worked out in previous studies. At the time of withdrawal, endpoint ratings will be made which include the full termination assessment battery.

Termination and post treatment assessment: At the end of the 12-week treatment period, all participants will be re-interviewed by the research assistant, who will complete post treatment ratings. Access to the CBT4CBT-COPES program will be terminated; however, participants in all conditions will be strongly encouraged to continue in agonist treatment at Liberation clinics.

Follow-up: Follow-up interviews will be conducted 1, 3, and 6 months after termination (the investigators find the one-month follow-up strengthens the relationship with the research staff and results in higher rates of follow-up). Follow-up interviews will include the full post-treatment battery, including assessment of utilization of other treatments and services. The investigators will attempt to follow all participants in the intention to treat sample, regardless of their retention in treatment, using strategies that have been successful in multiple previous studies. These include: (a) thorough explanation at the initial consent interview of the importance of follow-ups, (b) requiring that each participant provide at least 2 verified locators with knowledge of their whereabouts throughout follow-up, (c) use of multiple sources and locators to track participants, and (d) participant payment of $35 for each completed follow-up interview, with additional incentives for completing interviews on time and for completing consecutive follow-up interviews. Using these procedures, the investigators current rate of follow-up approaches 90-95% across studies for intention-to-treat analyses. For those who drop-out and cannot be re-engaged, the investigators will ask participants to complete a brief survey exploring their reasons for dropping out.

Rationale for study length: Given the 3-year limit for the R33 phase, in order to recruit a sample size for adequate power, the investigators decided to evaluate primary outcomes at 3 months, with an additional 6 months of follow-up (9-month total study period). This will allow the investigators to evaluate retention in OAT at the 6-month point. This should be adequate, as the bulk of attrition in OAT tends to occur earlier in treatment. Three months will allow for adequate exposure to the CBT4CBT-IMPACT intervention for those assigned to that condition; the additional 6 months of follow-up will allow evaluation of durability of treatment effects, and importantly, pain symptoms and use of health services for an adequate period.

Rationale for design: While a 3- or 4-cell design would allow for the integrated CBT4CBT-IMPACT intervention to be tested against either CBT4CBT or IMPACT alone, because of the 3 year time limit for the R33 phase and the emphasis on adequate power for the trial, the investigators decided the two-cell design would allow the investigators to determine if the integrated approach improves adherence and pain outcomes over standard OAT treatment in an adequately powered trial. If determined to be effective here, subsequent studies could evaluate the efficacy of the integrated approach relative to CBT4CBT or IMPACT alone, which would also allow for detailed evaluation of mechanism. Recruiting from a large specialty program will allow the investigators to recruit adequate numbers of both buprenorphine and methadone patients and hence enable some comparisons; this would be difficult in most primary care clinics. The Liberation evening clinic is similar to many office-based buprenorphine settings.

Treatments Standard care treatment as usual (TAU): Participants randomized to this condition will receive treatment-as-usual for the buprenorphine and methadone programs at Liberation Clinics, which includes regular medication management by the clinic physician, regular individual and group sessions and access to other services as needed. The investigators have worked closely with Liberation Clinics for over 20 years; the investigators selected this program because they are high-quality, well-managed programs which have supported multiple clinical research programs (including both Yale and CTN multi-site randomized trials of behavioral and pharmacologic approaches. All patients will also have access to counseling delivered onsite by highly experienced masters-level counselors employed at Liberation Clinics. Methadone and buprenorphine adherence will be monitored closely (via Timeline FollowBack as well as daily methadone visits, verification of buprenorphine prescriptions and counts, and evidence of buprenorphine/methadone in weekly urine toxicology screens). Utilization of all services (including counseling, medical care, ED visits, legal services, pharmacological and non-pharmacologic treatments for pain, etc.) will be monitored closely throughout the trial and through follow-up, in all conditions, using the PACC-SAT .

CBT4CBT-IMPACT. Participants assigned to this condition will receive standard agonist treatment but also receive access to CBT4CBT-IMPACT. At the time of randomization, participants will be given a username and asked to select a password to access the CBT4CBT-IMPACT website. The research staff will work with each participant to determine when, where, and how they will access the program (although participants will be free to access the program in a private area at the clinic as well). For the first session, research staff will guide the patient through the program to assure they are comfortable using the program and answer any questions they might have. Participants will be asked to spend at least one hour per week working with the program, either at the clinic or outside of the clinic (e.g. at their home). Participants will be asked to complete all 9 modules over the course of the 12-week study treatment period, repeating any modules, or sections, as they desire. At the start of each session, the study staff reviews the modules that the user has completed and directs users to either complete modules they have started or access new ones. The program tracks, for each participant, time logged onto the program, modules accessed, session progress, completion of practice exercises, and learning of CBT principles through multiple choice tests at the end of each module. Participants randomized to this condition will also be provided with a pocket pedometer to facilitate their participation in the walking portion of the treatment. Study staff will measure each participant's stride length, adjust the pedometer stride length setting accordingly, and provide a brief demonstration of pedometer use. Pedometers will record only steps.

Daily texts with a link for survey: Following randomization to CBT4CBT-IMPACT, participants will undergo daily assessment via text of pain intensity, pain interference, pedometer-measured step counts, sleep quality, sleep duration, and craving for seven days to establish a baseline of function for the purposes of treatment and providing regular feedback using questions derived from validated measures and used in our prior trials. After the baseline period, participants will continue to receive daily texts for the duration of the treatment. During treatment, two additional questions regarding practice of the treatment skills and progress toward the weekly meaningful activity goal will be included. Patient-reported data collected on the daily texts with link to a survey will form the basis for regular feedback, which will be tracked and viewed in graphical form from the patient dashboard of the program. Participants will receive texts with a link to a survey each day at a time pre-selected by the patient. Surveys will be no longer than 2 minutes in duration.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 18 years of age or older
* Meet DSM-5 criteria for OUD
* Enrolled in methadone or buprenorphine treatment at Liberation
* Have at least moderate-intensity chronic pain as indicated by a score of ≥ 4 over the past week on the 0-10 Numerical Rating Scale
* Have pain on at least half of the days of the prior six months (indicating chronicity);
* Self-reported ability to walk at least one block (for the exercise component of CBT4CBT-COPES

Exclusion Criteria:

* Inability to read, write, and speak English at a third grade level (for reading informed consent)
* Untreated or inadequately treated bipolar or psychotic disorder or current suicide risk as identified by Structured Clinical Interview for DSM-5 (SCID-5)
* Life threatening health conditions that would impede participation (e.g., end stage renal failure, malignant cancer requiring chemotherapy excluding melanoma)
* Planned surgical treatment related to pain
* Pending legal action or planned relocation that makes it unlikely they would be able to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Adherence to opioid agonist treatment (OAT) | Up to 36 weeks
  Adherence to opioid agonist treatment (OAT) will be verified by TimeLine Follow-back and clinic medical records of dates of medication taken, prescriptions filled and pick up. Individual adherence will be measured as a count. It will be measured at Weeks 12, 16, 24 and 36 weeks.
Change in PROMIS 6-item Pain Interference Short Form | Up to 36 weeks
  Pain interference is measured using the PROMIS 6-item Pain Interference Short Form. The range on the PROMIS Pain Form is 0 - 24, where 24 is the highest score and highest measure of pain. It will be measured at Weeks 12, 16, 24 and 36 weeks.

SECONDARY OUTCOMES:
Drug Use | Up to 36 weeks
  Opioid and other drug use will be assessed in participants using Urine toxicology screens and Timeline Follow-Back. Individual drug use will be measured as a count. It will be measured at Weeks 12, 16, 24 and 36 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Heapy, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Liberation Programs, Bridgeport, Connecticut
  - Connecticut Counseling Center, Danbury, Connecticut
  - Connecticut Counseling Centers, Waterbury, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacLean RR, Ankawi B, Driscoll MA, Gordon MA, Frankforter TL, Nich C, Szollosy SK, Loya JM, Brito L, Ribeiro MIP, Edmond SN, Becker WC, Martino S, Sofuoglu M, Heapy AA. Efficacy of Integrating the Management of Pain and Addiction via Collaborative Treatment (IMPACT) in Individuals With Chronic Pain and Opioid Use Disorder: Protocol for a Randomized Clinical Trial of a Digital Cognitive Behavioral Treatment. JMIR Res Protoc. 2024 Mar 20;13:e54342. doi: 10.2196/54342. PMID 38506917